CLINICAL TRIAL: NCT03291184
Title: Is Postoperative Residual Curarisation Still an Issue at the Moment of Weaning of the ICU Patient Following Cardiac Surgery?
Brief Title: Postoperative Residual Paralysis After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Guy CAMMU, MD, PhD, Staff Anesthesiologist, Onze Lieve Vrouw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: EN_GC_2017
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Residual Curarization
Keywords: neuromuscular blockade; neuromuscular monitoring
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Intervention Model Description: Patients admitted to the ICU after elective cardiac surgery and ready for weaning from the ventilator.
Who Masked: Participant, Investigator
Masking Description: The participant will still be under sedation at the moment of measuring neuromuscular blockade. The care provider will perform measurements, while the investigator is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: peripheral neuromuscular monitor — Residual paralysis can only be measured by neuromuscular transmission monitoring of a peripheral nerve, typically the ulnar nerve innervating the adductor pollicis muscle.

SUMMARY:
The main objective of this study is to describe the incidence of postoperative residual paralysis (mean train-of-four <90%) when weaning from the ventilator in patients admitted to the Intensive Care Unit (ICU) after elective cardiac surgery. Train-of-four monitoring is a widely used term for the peripheral nerve stimulation used in neuromuscular blockade monitoring. When the patient is ready for weaning from the ventilator, an ICU doctor will perform a measurement of the train-of-four at the thumb with a neuromuscular transmission monitor. Every value below 90% will be considered as residual paralysis and treated appropriately by means of a reversal agent.

DETAILED DESCRIPTION:
Postoperatively, in the ICU, readiness-for-weaning is based on ICU doctor-nurse-driven institutional weaning guidelines: 6 hours after arrival in the ICU, a patient who is normothermic, hemodynamically stable, has normal blood gasses and absence of residual bleeding. The ICU nurse caring for the patient will start weaning the patient from the ventilator, following these departmental guidelines.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the ICU after elective cardiac surgery

Exclusion Criteria:

* emergency cardiac surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-03-08 (Actual)

PRIMARY OUTCOMES:
postoperative residual curarisation | 6 hours after arrival in the ICU
  mean train-of-four <90% as measured by neuromuscular blockade monitoring

CONTACTS AND LOCATIONS:
Overall Officials: GUY CAMMU, Principal Investigator — Onze-Lieve-Vrouw Ziekenhuis Aalst, Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cammu G. How rational is muscle relaxation during cardiac surgery? Acta Anaesthesiol Belg. 2007;58(1):7-14. PMID 17486918
- [Background] Videira RL, Vieira JE. What rules of thumb do clinicians use to decide whether to antagonize nondepolarizing neuromuscular blocking drugs? Anesth Analg. 2011 Nov;113(5):1192-6. doi: 10.1213/ANE.0b013e31822c986e. Epub 2011 Aug 24. PMID 21865491
- [Background] Rudis MI, Guslits BG, Zarowitz BJ. Technical and interpretive problems of peripheral nerve stimulation in monitoring neuromuscular blockade in the intensive care unit. Ann Pharmacother. 1996 Feb;30(2):165-72. doi: 10.1177/106002809603000211. PMID 8835051